CLINICAL TRIAL: NCT01273402
Title: Pretargeted Radioimmunotherapy of Colorectal Cancer: A Phase I Study to Determine Dose-limiting Toxicity and Maximum Tolerated Dose of an Anti-CEACAM5 bsMAb-pretargeted 90Y-hapten-peptide
Brief Title: Study of TF2 Carcinoembryonic Antigen (CEA) Antibody in Patients With Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: A new study is being designed. No patients were enrolled.
Sponsor: Gilead Sciences (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Robert Sharkey, PhD, Garden State Cancer Center/Center for Molecular Medicine and Immunology
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-072-09 (NCI 5R01CA107088-04); 5R01CA107088-04 (NIH)
Record Dates: First submitted 2011-01-05; First posted 2011-01-10 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; TF2 (Recombinant, humanized Tri-Fab bsMAb composed of 2 humanized MN-14 anti-CEA Fab x and one 679 anti-HSG Fab); IMP288 (DOTA-di-HSG hapten-peptide for 111In/90Y labeling)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — DOTA-tyrosyl-lysyl(histaminyl-succinyl-glycyl)-glutamyl-lysyl(histaminyl-succinyl-glycyl)amide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TF2 and IMP288 (Experimental): TF2 will be administered at least 4 days before the radiolabeled IMP-288.
  Interventions: Drug: TF2/IMP288

INTERVENTIONS:
Drug: TF2/IMP288 — TF2 is administered 4 days prior to radiolabeled IMP288. Each are given weekly for 2 weeks.
  Other Names: TF2; IMP288; bi-specific antibodies; pre-targeted antibodies

SUMMARY:
This study is being done to select an appropriate TF2 bsMAb dose suitable for pretargeting the 111In/90Y-labeled hapten-peptide (IMP-288). Eligible patients will receive a fixed dose of 90Y-IMP-288 4 days after the TF2 antibody injection. Two different dose levels of TF2 will be studied in the first part.

Once an appropriate TF2 dose is selected based on information learned from the first 2 dose levels, patients will be enrolled onto several different increasing dose levels of 90Y-IMP-288.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, >18 years of age.
* documented histologic or cytologic diagnosis of metastatic (Stage IV) colorectal cancer.
* must have at least one confirmed and measurable tumor lesion (a confirmed tumor site is one in which either biopsy-proven evidence of disease or progressive growth has been radiographically observed).
* Patients must have failed standard therapy or for whom no standard therapy exists.
* Patients must have a Karnofsky performance status of ≥ 70% (or equivalent ECOG 0-1) and an expected survival of ≥ 3 months.
* Patients who previously received a chimeric, CDR-grafted (humanized), or human IgG will be eligible provided pre-study evaluations demonstrate no significant anti-antibody reactivity with TF2.
* Hematologic parameters: WBC counts must be ≥ 3000/mm3, granulocytes

  * 1500/mm3, and platelets ≥ 100,000/m3.
* Non-hematologic parameters: Patients without liver metastases must have bilirubin ≤ 1.5 institutional upper limit of normal (IULN), whereas bilirubin in patients with known liver metastases must be <2.5-times the IULN. AST/ALT must not be >2.5 times IULN.
* At least 2 weeks beyond corticosteroids, except low doses (i.e., 20 mg/day of prednisone or equivalent) to treat nausea or other illness such as rheumatoid arthritis.
* Patients able to understand and give written informed consent. Informed consent must be obtained prior to baseline studies for enrollment purposes.

Exclusion Criteria:

* Women who are pregnant or lactating. Women of childbearing potential and fertile men will be informed as to the potential risk of procreation while participating in this trial and will be advised that they must use effective contraception during and for a period of 3 months.
* Patients with plasma CEA >1000 ng/mL or lesions exceeding 10 cm in diameter.
* Patients with severe anorexia or other gastrointestinal-related symptomatology (e.g., nausea, vomiting).
* Patients with known HIV or hepatitis B or C.
* Patients with an active second primary malignancy at the time of study entry, with the exception of carcinoma in situ of the cervix.
* Patients with known metastatic disease to the central nervous system.
* Patients with evidence of bone marrow metastases. Screening only required for patients with suspicion of metastases. Patients with ≥ 25% bone marrow involvement are excluded.
* Patients who are, in the opinion of the investigator, unable to comply with the protocol requirements.
* Institutionalized subjects (e.g., prisons, psychiatric facilities).
* Known history of active coronary artery disease, unstable angina, myocardial infarction, or congestive heart failure present within 6 months or cardiac arrhythmia requiring anti-arrhythmia therapy.
* Known autoimmune disease or presence of autoimmune phenomena (except rheumatoid arthritis requiring only low dose maintenance corticosteroids); or infection requiring intravenous antibiotic use within 1 week.
* Known history of active COPD, or other moderate-to-severe respiratory illness present within 6 months.
* Patients who are diabetic and/or have high blood pressure are at a higher risk for developing late-stage renal failure. While these patients will not be specifically excluded, physician-investigators must carefully discuss the associated late risks to these patients.
* Patients must be at least 4 weeks beyond prior chemotherapy, surgery, radiotherapy to an index lesion, or experimental therapy (i.e., drugs, biologicals, procedures) and meet all eligibility criteria.
* Patients who received a treatment containing a nitrosourea compound will not be enrolled for at least 6 weeks after the end of that treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Determine the number of adverse events | Safety will be measured routinely during the 3 weeks of administration and afterwards during follow-up for up to 5 years
  Safety will be assessed by determing the number of participants with Adverse Events as a Measure of Safety and Tolerability.

SECONDARY OUTCOMES:
Efficacy will be evaluating using CT scans and possibly PET imaging. | Efficacy will be measured at 4 and 8 weeks after treatment and every 3 months for up to 2 years.
  CT scans will primarily be used to assess tumor response and to assess the change in tumor size from baseline for up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sharkey, PhD, Principal Investigator — Garden State Cancer Center/Center for Molecular Medicine and Immunology
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Schoffelen R, van der Graaf WT, Franssen G, Sharkey RM, Goldenberg DM, McBride WJ, Rossi EA, Eek A, Oyen WJ, Boerman OC. Pretargeted 177Lu radioimmunotherapy of carcinoembryonic antigen-expressing human colonic tumors in mice. J Nucl Med. 2010 Nov;51(11):1780-7. doi: 10.2967/jnumed.110.079376. PMID 21051650
- [Background] Sharkey RM, Rossi EA, McBride WJ, Chang CH, Goldenberg DM. Recombinant bispecific monoclonal antibodies prepared by the dock-and-lock strategy for pretargeted radioimmunotherapy. Semin Nucl Med. 2010 May;40(3):190-203. doi: 10.1053/j.semnuclmed.2009.12.002. PMID 20350628
- [Background] Chatal JF, Campion L, Kraeber-Bodere F, Bardet S, Vuillez JP, Charbonnel B, Rohmer V, Chang CH, Sharkey RM, Goldenberg DM, Barbet J; French Endocrine Tumor Group. Survival improvement in patients with medullary thyroid carcinoma who undergo pretargeted anti-carcinoembryonic-antigen radioimmunotherapy: a collaborative study with the French Endocrine Tumor Group. J Clin Oncol. 2006 Apr 10;24(11):1705-11. doi: 10.1200/JCO.2005.04.4917. Epub 2006 Mar 20. PMID 16549819
- [Background] Kraeber-Bodere F, Rousseau C, Bodet-Milin C, Ferrer L, Faivre-Chauvet A, Campion L, Vuillez JP, Devillers A, Chang CH, Goldenberg DM, Chatal JF, Barbet J. Targeting, toxicity, and efficacy of 2-step, pretargeted radioimmunotherapy using a chimeric bispecific antibody and 131I-labeled bivalent hapten in a phase I optimization clinical trial. J Nucl Med. 2006 Feb;47(2):247-55. PMID 16455630
- [Background] Kraeber-Bodere F, Faivre-Chauvet A, Ferrer L, Vuillez JP, Brard PY, Rousseau C, Resche I, Devillers A, Laffont S, Bardies M, Chang K, Sharkey RM, Goldenberg DM, Chatal JF, Barbet J. Pharmacokinetics and dosimetry studies for optimization of anti-carcinoembryonic antigen x anti-hapten bispecific antibody-mediated pretargeting of Iodine-131-labeled hapten in a phase I radioimmunotherapy trial. Clin Cancer Res. 2003 Sep 1;9(10 Pt 2):3973S-81S. PMID 14506196
- [Background] Kraeber-Bodere F, Goldenberg DM, Chatal JF, Barbet J. Pretargeted radioimmunotherapy in the treatment of metastatic medullary thyroid cancer. Curr Oncol. 2009 Sep;16(5):3-8. doi: 10.3747/co.v16i5.464. No abstract available. PMID 19862356
- [Background] Goldenberg DM, Chatal JF, Barbet J, Boerman O, Sharkey RM. Cancer Imaging and Therapy with Bispecific Antibody Pretargeting. Update Cancer Ther. 2007 Mar;2(1):19-31. doi: 10.1016/j.uct.2007.04.003. PMID 18311322
- [Background] Goldenberg DM, Sharkey RM, Paganelli G, Barbet J, Chatal JF. Antibody pretargeting advances cancer radioimmunodetection and radioimmunotherapy. J Clin Oncol. 2006 Feb 10;24(5):823-34. doi: 10.1200/JCO.2005.03.8471. Epub 2005 Dec 27. PMID 16380412